CLINICAL TRIAL: NCT04762082
Title: A Single Dose Randomized Five-Way Crossover Pharmacokinetics (PK) Study of Tadalafil Semi-Chewable (Gummy) Formulations in Healthy Volunteers
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Gummy Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: P-002-2020
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Eligible subjects will receive a single oral dose of one of five treatments (Treatments A, B, C, D or E) in five separate periods in a randomly assigned sequence, with each treatment separated by an approximate 5-day washout period. In each study period, dosing will occur in the morning after an overnight fast of at least 10 hours.
  All doses will be administered under fasted conditions except for Treatment C, when tadalafil gummy 10 mg will be administered after consumption of a high-calorie, high-fat breakfast.
  All doses will be administered with approximately 240 mL of room temperature water except for Treatment D, when tadalafil gummy 10 mg dose will be administered without water.
  All doses of tadalafil gummy 10 mg will be chewed before swallowing except for Treatment E, when subjects will be instructed to swallow the dose whole.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Treatment A: Test (Experimental): Single oral dose of tadalafil gummy 10 mg, chewed, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: Tadalafil 10 MG
- Treatment B: Reference (Active Comparator): Single oral dose of tadalafil oral tablets 10 mg, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: Tadalafil 10 MG
- Treatment C: Test (Experimental): Single oral dose of tadalafil gummy 10 mg, chewed, administered with approximately 240 mL of room temperature water, under fed conditions
  Interventions: Drug: Tadalafil 10 MG
- Treatment D: Test (Experimental): Single oral dose of tadalafil gummy 10 mg, chewed, administered with no water, under fasted conditions
  Interventions: Drug: Tadalafil 10 MG
- Treatment E: Test (Experimental): Single oral dose of tadalafil gummy 10 mg, swallowed whole, administered with approximately 240 mL of room temperature water, under fasted conditions
  Interventions: Drug: Tadalafil 10 MG

INTERVENTIONS:
Drug: Tadalafil 10 MG — comparison of tadalafil gummy 10mg and tadalafil oral tablet 10mg

SUMMARY:
This is a randomized, open-label, single-dose, five-period crossover, relative bioavailability study to evaluate tadalafil gummy 10mg and tadalafil oral tablets 10mg in healthy volunteers

DETAILED DESCRIPTION:
This is an open-label, single dose, randomized, five-period, crossover design study to evaluate the relative bioavailability of a single oral dose of tadalafil gummy 10 mg (Test) and tadalafil oral tablets 10 mg (Reference) under fasted conditions in healthy adult male and female subjects, and the impact on the bioavailability of tadalafil gummy sugar free 10 mg when administered with food, when administered with or without water, and when chewed or swallowed whole.

Each subject will receive tadalafil gummy (10 mg) or tadalafil tablet and thereby will be his/hers own control.

ELIGIBILITY:
Inclusion Criteria:

* male 19-65 years of age;
* Available to participate for the planned duration of the study;
* Able and willing to complete the informed consent process;
* Agree to have blood samples collected and stored for the study;
* Agree not to use approved or experimental benign prostatic hyperplasia or erectile dysfunction treatments anytime during the course of the study;
* Have not taken finasteride or dutasteride therapy, any other lower urinary tract symptom (LUTS) therapy or phosphodiesterase type 5 (PDE5) inhibitors for specified duration of time prior to the study;
* Have not taken nitrates, alpha blockers, antihypertensives, alcohol, CYP3A4 inhibitors and CYP3A4 inducers for a specified duration of time prior to the study;
* Have a prostate specific antigen (PSA) score within acceptable range defined for study or negative biopsy of the prostate for cancer within 12 months of the study.

Exclusion Criteria:

* A condition in which repeated blood draws poses more than minimal risk for the subject such as hemophilia, other severe coagulation disorders or significantly impaired venous access;
* A condition that requires active medical intervention or monitoring to avert serious danger to the subject's health or well-being;
* subjects with dentures, partial dentures or braces, subjects with swallowing disorders and subjects who abuse drugs, alcohol or tobacco;
* Currently taking nitrates or nitro compounds, alpha blockers, antihypertensives, alcohol, CYP3A4 inhibitors, CYP3A4 inducers;
* Currently taking any medicines known to conflict with tadalafil;
* History of urinary retention or lower urinary tract (bladder) stones 6 months before the start of the study;
* History of bladder outlet obstruction or urethral obstruction due to stricture, valves, sclerosis, or tumor;
* History of diabetes;
* History of cardiac conditions including angina requiring certain treatment with nitrates, heart disease or coronary conditions including myocardial infarction, bypass surgery, angioplasty or stent placement for a specified time before starting the study;
* Certain neurological conditions associated with bladder problems or injuries to the brain or spinal cord within a specified time before starting the study.

Ages: 19 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
maximum plasma cetirizine concentration (Cmax) | 96 hours
  PK blood samples to measure plasma concentrations of tadalafil will be collected by direct venipuncture or by use of an indwelling cannula. Blood will be collected into tubes containing K2EDTA for determination of plasma tadalafil concentration at time 0 (within 60 minutes pre-dose), 10, 20 minute post-dose and 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 24, 48, 72 and 96 hours post-dose. Plasma tadalafil concentrations will be listed at each time point by subject and summarized by treatment at each time point using descriptive statistics (n, mean, standard deviation (SD), Coefficient of variation (CV%), median, minimum and maximum values). Pharmacokinetic calculations will be performed based on actual time of blood sample collection, using non-compartmental methods with Phoenix WinNonlin Version 8.1 (Certara USA, Inc., Princeton, New Jersey, USA). Plots of mean concentrations of plasma tadalafil versus time will be generated and Cmax will be generated from the plot.
area under the plasma drug concentration versus time curve (AUC) | 96 hours
  AUC will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ). AUC will be calculated to the last measurable observation (AUC0-t) and extrapolated to infinity (AUC0 ∞).

SECONDARY OUTCOMES:
time to Cmax (Tmax) | 96 hours
  Tmax will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).
elimination half-life (t½) | 96 hours
  t½ will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).
terminal elimination rate constant (Kel). | 96 hours
  Kel will be determined using non-compartmental analysis methods (Phoenix WinNonlin software, version 8.1 or higher, Certara USA Inc., Princeton, NJ).

IPD SHARING:
Plan to Share IPD: No